CLINICAL TRIAL: NCT00753662
Title: Phase 2 (Feasibility) Study of Transcranial Magnetic Stimulation as Additional Therapy to Drug Treatment in Patients With Alzheimer's Disease
Brief Title: Deep Transcranial Magnetic Stimulation in Patients With Alzheimer's Disease
Acronym: TMS in AD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Brainsway (Industry)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Dr. Alissa Ash, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TASMC-08-AA-0397-CTIL
Record Dates: First submitted 2008-09-14; First posted 2008-09-16 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Alzheimer's Disease
Keywords: TMS AD H2 coil
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 15 patients in group 1 will be treated with 1Hz frequency
  Interventions: Device: 1Hz TMS with H2 coil
- 2 (Active Comparator): 15 patients in group 2 will be treated with 1Hz frequency 10Hz
  Interventions: Device: 10Hz TMS with H2 coil to prefrontal and parieto-temporal cortex
- 3 (Sham Comparator): 15 patients in group 3 will be treated with SHAM (1Hz/10Hz)
  Interventions: Device: SHAM TMS with H2 coil

INTERVENTIONS:
Device: 1Hz TMS with H2 coil — 1Hz TMS with H2 coil to prefrontal and parieto-temporal cortex
  Arms: 1
Device: 10Hz TMS with H2 coil to prefrontal and parieto-temporal cortex — 10Hz TMS with H2 coil to prefrontal and parieto-temporal cortex
  Other Names: 10Hz TMS with H2 coil
  Arms: 2
Device: SHAM TMS with H2 coil — SHAM TMS with H2 coil to prefrontal and parieto-temporal cortex
  Arms: 3

SUMMARY:
The primary objective of this trial is to assess the ability of Transcranial Magnetic Stimulation with H2 coil to prefrontal and parieto-temporal cortex to improve cognitive performance in patients with Alzheimer's disease which received drug treatment. This study is a single-center, double-blind 4 months duration trial.

DETAILED DESCRIPTION:
Primary outcome measure: ADAS-COG (time frame baseline, 2 months, 4 months) Secondary outcome measure: CGI-C, Neuropsychological computerized test (Mindstream), FAB,ADL, Beck Depression Inventory-time frame baseline,1 month (visit 12) 2 months (visit 16), 4 months (visit 17).

Estimated enrollment: 45 patients Estimated Study start Date: November 2008 Estimated Study Completion date: November 2012 Number of arms: 3 Interventions details: H2 coil device for Transcranial Magnetic Stimulation with MAGSTIM to prefrontal and parieto-temporal regions bilaterally with frequency 10Hz in one arm, 1Hz in the second arm, and sham-stimulation with frequency 10Hz/1Hz in third arm.

Ages: 50-80 Genders: both

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent will be obtained
* diagnostic evidence of probable AD consistent with DSM IV
* stable treatment with Acetylcholine-Esterase Inhibitors or/and Memantine for 5 weeks prior to screening
* stable dose treatment with other drugs
* MMSE <25

Exclusion Criteria:

* Patients with neurological or psychiatric disorders that affect cognition but are distinguishable from AD
* Patients who are unwilling or unable to fulfill the requirements of the study
* Severe personality disorder
* Malignant or untreated Hypertension
* History of Epilepsy
* History of Head trauma
* Metal implant in head, cardiac pacemaker, medical pump
* Drug or alcohol addiction
* Involvement in any other clinical trial during the preceding 3 month
* Patient who are unwilling or unable to give Informed Consent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
ADAS-COG | Baseline, 1 month (visit 12), 2 months (visit 16), 4 months (visit 17)

SECONDARY OUTCOMES:
CGI-C, Neuropsychological computerized test (Mindstream),CGI-C,FAB,ADL, Beck Depression Inventory. | Baseline, 1 month (visit 12), 2 months (visit 16), 4 months (visit 17)

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Ash, Dr., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Neurology Department, Tel Aviv, Israel